CLINICAL TRIAL: NCT05439941
Title: A Long-Term Extension Trial in Participants With Atopic Dermatitis Who Participated in Previous Phase 2 And 3 EDP1815 Trials
Brief Title: A Long-Term Extension Trial in Participants With Atopic Dermatitis Who Participated in Previous EDP1815 Trials
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Parent Study (NCT05121480) did not meet the primary endpoint.
Sponsor: Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDP1815-208; 2022-000284-48 (EudraCT Number)
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Results first posted 2023-09-07 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-08

CONDITIONS: Atopic Dermatitis
Keywords: Mild Atopic Dermatitis; Moderate Atopic Dermatitis; Severe Atopic Dermatitis; Mild Eczema; Moderate Eczema; Severe Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Intervention Model Description: Open Label Extension Study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (1.6x10^11 total cells of EDP1815, 2 capsules once daily) (Experimental): EDP1815-207 Cohort 1 participants will receive 1.6x10^11 total cells of EDP1815 in EDP1815-208 administered as 2 capsules once daily. (Group 1)
  Interventions: Drug: EDP1815
- Group 2 (6.4x10^11 total cells of EDP1815, 2 capsules once daily) (Experimental): EDP1815-207 Cohort 2 participants will receive 6.4x10^11 total cells of EDP1815 in EDP1815-208 administered as 2 capsules once daily. (Group 2)
  Interventions: Drug: EDP1815
- Group 3 (8.0x10^10 total cells of EDP1815, 1 capsule once daily) (Experimental): EDP1815-207 Cohort 4 participants will receive 8.0x10^10 total cells of EDP1815 in EDP1815-208 administered as 1 capsule once daily. (Group 3)
  Interventions: Drug: EDP1815

INTERVENTIONS:
Drug: EDP1815 — EDP1815 is an orally administered, pharmaceutical preparation of a single strain of bacteria
  Other Names: Prevotella histicola

SUMMARY:
This is an Open-Label Extension (OLE) study to evaluate the long-term safety, tolerability, and efficacy of EDP1815 in participants with mild, moderate, and severe atopic dermatitis who have completed the treatment period of a prior clinical study ("parent study") with EDP1815.

The current parent study of this protocol is the EDP1815-207 study; A Phase 2, Multicenter, Double-Blind, Placebo-Controlled, Multiple-Cohort Study Investigating the Effect of EDP1815 in Participants for the Treatment of Mild, Moderate and Severe Atopic Dermatitis.

DETAILED DESCRIPTION:
Atopic dermatitis (atopic eczema) is a very common type of skin disease. It typically causes red, dry, and itchy skin and may have a significant impact on quality of life. Rashes may appear on the arms and behind the knees, or anywhere else on the body. While there are existing therapies, there is currently no cure for atopic dermatitis.

This study is an Open Label Extension (OLE) study to the first parent study; i.e., the EDP1815-207 study (NCT05121480). The total number of participants will be dependent on the number of participants who elect and are eligible to participate in the Open Label Extension study following participation in EDP1815-207.

All participants in this study will be treated with EDP1815, regardless of the treatment assignment in the EDP1815-207 study. There will be no placebo drug administered in this study. To minimize bias, during dosing in EDP1815-208, investigators and participants will continue to be blinded to participants' treatment allocation in the parent study whilst it is ongoing. Participants in this study will be treated with EDP1815 for up to 36 weeks, followed by a follow-up visit at approximately 4 weeks after the end of treatment.

The maximum study duration is up to 40 weeks for all participants. The participants may move directly from the parent study into the open label treatment phase without a break in study treatment, or within 7 days of completing the treatment period of the parent study. If the participants move directly into this study without a break in treatment from the parent study, the Day -1 visit should be performed at the same time as the end of treatment visit of the parent study.

The primary endpoint of safety and tolerability will be measured using the incidence and rate per 100 patient-years of treatment-emergent adverse events during the 36-week treatment period and the 4-week follow-up period of this study; and during the treatment period of this study and the parent study. TEAEs will be defined as all events starting after first dose of study drug, and on or before 28 days after last dose for each participant. All TEAEs will be included in the assessments of incidences and rates, regardless of compliance with study medication, use of other medications or deviations from the study protocol.

The secondary endpoint of efficacy will be measured using the Eczema Area and Severity Index (EASI) Score. Additionally, the Investigator's Global Assessment (IGA), percentage of Body Surface Area (BSA), Product of the IGA and BSA (IGA*BSA), the SCORing Atopic Dermatitis (SCORAD), the Dermatology Life Quality Index (DLQI), the Peak Pruritus Numerical Rating Scale (PP-NRS), the Sleep Disturbance Numerical Rating Scale (SD-NRS), the Patient Oriented Eczema Measure (POEM) and the Atopic Dermatitis Control Tool (ADCT) will also be measured throughout the study. The number of courses of treatment with rescue therapies; and with antibiotic treatment due to skin infection, per participant, will also be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Must have provided informed consent.
2. Must have completed the treatment period in a parent study of EDP1815 in atopic dermatitis and complied with the parent protocol.
3. Must agree to use emollients.
4. Must continue to follow contraception criteria.

Exclusion Criteria:

1. Participants who are currently enrolled in another investigational drug study or plans to receive another investigational drug during this study.
2. Have any other conditions, which would make the participant unsuitable for inclusion or could interfere with the participant participating in or completing the study.
3. Use of phototherapy, a biologic agent, or a systemic immunosuppressive agent that could affect AD, including systemic corticosteroids, within 7 days prior to Day -1, unless used as a rescue treatment as part of the parent study protocol.
4. Use of topical atopic dermatitis therapies, including topical corticosteroids, topical calcineurin inhibitors, topical PDE-4 inhibitors, and topical JAK inhibitors, within 7 days prior to enrolling in the study, unless used as a rescue treatment as part of the EDP1815-207 protocol.
5. Has received live or live-attenuated vaccination prior to enrollment or intends to have such a vaccination during the study.
6. Hypersensitivity to P histicola or to any of the excipients.
7. Unwillingness to comply with study procedures, including follow-up, as specified by this protocol, or unwillingness to cooperate fully with the Investigator.

Ages: 18 Years to 76 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Maslin, MD, Study Director — Evelo Biosciences; Ben Ehst, PhD, Principal Investigator — Oregon Medical Research Center
Locations (54):
- United States (24):
  - USA-131, Birmingham, Alabama
  - USA 112, Fountain Valley, California
  - USA 123, Fremont, California
  - USA -101, Fort Lauderdale, Florida
  - USA-124, Jacksonville, Florida
  - USA-108, Miami, Florida
  - USA-120, Miami, Florida
  - USA-105, Miramar, Florida
  - USA-102, Orlando, Florida
  - USA-115, Sweetwater, Florida
  - USA-106, Tampa, Florida
  - USA-126, Tampa, Florida
  - USA-111, Clarksville, Indiana
  - USA-116, Louisville, Kentucky
  - USA-119, Baton Rouge, Louisiana
  - USA-109, Metairie, Louisiana
  - USA-125, Silver Spring, Maryland
  - USA-121, Columbus, Ohio
  - USA-128, Concord, Ohio
  - USA-104, Portland, Oregon
  - USA-127, Memphis, Tennessee
  - USA-117, Frisco, Texas
  - USA-110, Pflugerville, Texas
  - USA-113, Bellevue, Washington
- Australia (4):
  - AUS-102, Carlton
  - AUS-104, Kogarah
  - AUS-101, Melbourne
  - AUS-106, Woolloongabba
- Bulgaria (4):
  - BGR-105, Pleven
  - BGR-104, Sevlievo
  - BGR-101, Sofia
  - BGR-103, Sofia
- Canada (9):
  - CAN-109, Barrie
  - CAN-108, Edmonton
  - CAN-105, Markham
  - CAN-104, Mississauga
  - CAN-101, Ottawa
  - CAN-107, Richmond Hill
  - CAN-103, Surrey
  - CAN-106, Waterloo
  - CAN-111, Winnipeg
- Germany (6):
  - DEU-105, Berlin
  - DEU-106, Erlangen
  - DEU-102, Frankfurt am Main
  - DEU-104, Gera
  - DEU-101, Hamburg
  - DEU-103, Heidelberg
- Poland (7):
  - POL-104, Gdansk
  - POL-106, Gdynia
  - POL-107, Katowice
  - POL-105, Lodz
  - POL-101, Lublin
  - POL-102, Warsaw
  - POL-103, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Participants with mild, moderate or severe Atopic Dermatitis who received 2 capsules (1.6 x 10^11 total cells) of EDP1815 (an orally administered, pharmaceutical preparation of a single strain of bacteria) once daily.
- Group 2: Participants with mild, moderate or severe Atopic Dermatitis who received 2 capsules (6.4 x 10^11 total cells) of EDP1815 (an orally administered, pharmaceutical preparation of a single strain of bacteria) once daily.
- Group 3: Participants with mild, moderate or severe Atopic Dermatitis who received 1 capsule (8.0 x 10^10 total cells) of EDP1815 (an orally administered, pharmaceutical preparation of a single strain of bacteria) once daily.
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3
Started | 104 | 102 | 79
Completed | 0 | 0 | 0
Not Completed | 104 | 102 | 79
Not completed — Lack of Efficacy | 8 | 5 | 3
Not completed — Treatment Failure | 0 | 1 | 0
Not completed — Adverse Event | 1 | 3 | 0
Not completed — Adverse Event - Parent Study | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 6 | 10
Not completed — Non-Compliance | 1 | 1 | 1
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Trial Termination by Sponsor | 78 | 83 | 65
Not completed — Other than Reasons Listed | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Total
Number analyzed (Participants) | 104 | 102 | 79 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.0 (16.28) | 40.6 (14.05) | 39.4 (14.66) | 40.0 (15.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 49 | 45 | 147
  Male | 51 | 53 | 34 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 4 | 13
  Not Hispanic or Latino | 97 | 98 | 74 | 269
  Unknown or Not Reported | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 12 | 10 | 33
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 7 | 9 | 10 | 26
  White | 81 | 77 | 56 | 214
  More than one race | 3 | 3 | 2 | 8
  Unknown or Not Reported | 1 | 1 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 19 | 22 | 20 | 61
  United States | 25 | 25 | 19 | 69
  Poland | 30 | 25 | 29 | 84
  Australia | 4 | 4 | 1 | 9
  Bulgaria | 18 | 16 | 7 | 41
  Germany | 8 | 10 | 3 | 21

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Rate Per 100 Patient-years of Treatment-emergent Adverse Events
Description: The long-term safety and tolerability of EDP1815 in the treatment of atopic dermatitis will be measured by evaluating the incidence and rate per 100 patient-years of treatment-emergent adverse events during the 36-week treatment period and the 4-week follow-up period of this study, and during the treatment period of this study and the relevant parent study.
Time Frame: 40 weeks
Population: No participants reached the Week 40 timepoint for inclusion in the analysis as the study was terminated (halted early) as Parent Study (NCT05121480) did not meet the primary endpoint.
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Percentage of Participants Achieving EASI-50
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following EASI endpoints:
  • Percentage of participants achieving EASI-50
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Achieving EASI-75
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following EASI endpoints:
  • Percentage of participants achieving EASI-75
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Percentage of Participants Achieving EASI-90
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following EASI endpoints:
  • Percentage of participants achieving EASI-90
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Mean Absolute Change From Baseline in EASI Score
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following EASI endpoints:
  • Mean absolute change from baseline in EASI Score
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Mean Percentage Change From Baseline in EASI Score
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following EASI endpoints:
  • Mean percentage change from baseline in EASI Score
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving IGA of 0 or 1 With a ≥2 Point Improvement From Baseline
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following IGA endpoints:
  • Percentage of participants achieving IGA of 0 or 1 with a ≥2 point improvement from baseline
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Percentage of Participants Achieving IGA of 0 or 1
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following IGA endpoints:
  • Percentage of participants achieving IGA of 0 or 1
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Percentage of Participants Achieving IGA of 0
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following IGA endpoints:
  • Percentage of participants achieving IGA of 0
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Mean Absolute Change From Baseline in IGA*BSA
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following IGA *BSA endpoints:
  • Mean absolute change from baseline in IGA*BSA
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Mean Percentage Change From Baseline in IGA*BSA
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following IGA *BSA endpoints:
  • Mean percentage change from baseline in IGA*BSA
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Mean Absolute Change From Baseline in BSA
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following IGA *BSA endpoints:
  • Mean absolute change from baseline in BSA
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Mean Percentage Change From Baseline in BSA
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following IGA *BSA endpoints:
  • Mean percentage change from baseline in BSA
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Percentage of Participants Achieving BSA-50
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following IGA *BSA endpoints:
  • Percentage of participants achieving BSA-50
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

15. Secondary Outcome: Percentage of Participants Achieving BSA-75
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following BSA endpoints:
  • Percentage of participants achieving BSA-75
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Percentage of Participants Achieving BSA Reduction to 3% or Less
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following IGA *BSA endpoints:
  • Percentage of participants achieving BSA reduction to 3% or less
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Mean Absolute Change From Baseline in SCORAD
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following SCORAD endpoints:
  • Mean absolute change from baseline in SCORAD
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

18. Secondary Outcome: Mean Percentage Change From Baseline in SCORAD
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following SCORAD endpoints:
  • Mean percentage change from baseline in SCORAD
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

19. Secondary Outcome: Percentage of Participants Achieving SCORAD-50
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following SCORAD endpoints:
  • Percentage of participants achieving SCORAD-50
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Percentage of Participants Achieving SCORAD-75
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following SCORAD endpoints:
  • Percentage of participants achieving SCORAD-75
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Mean Absolute Change From Baseline in DLQI
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following DLQI endpoints:
  • Mean absolute change from baseline in DLQI
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Mean Percentage Change From Baseline in DLQI
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following DLQI endpoints:
  • Mean percentage change from baseline in DLQI
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥4 in the DLQI, of Those With a Score of ≥4 at Baseline
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following DLQI endpoints:
  • Percentage of participants achieving a reduction of ≥4 in the DLQI, of those with a score of ≥4 at baseline
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Mean Absolute Change From Baseline in PP-NRS
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following PP-NRS endpoints:
  • Mean absolute change from baseline in PP-NRS
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥2 in the PP-NRS, of Those With a Score of ≥2 at Baseline
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following PP-NRS endpoints:
  • Percentage of participants achieving a reduction of ≥2 in the PP-NRS, of those with a score of ≥2 at baseline
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥4 in the PP-NRS, of Those With a Score of ≥4 at Baseline
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following PP-NRS endpoints:
  • Percentage of participants achieving a reduction of ≥4 in the PP-NRS, of those with a score of ≥4 at baseline
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Mean Absolute Change From Baseline in SD-NRS
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following SD-NRS endpoints:
  • Mean absolute change from baseline in SD-NRS
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥2 in the SD NRS, of Those With a Score of ≥2 at Baseline
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following SD-NRS endpoints:
  • Percentage of participants achieving a reduction of ≥2 in the SD NRS, of those with a score of ≥2 at baseline
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

29. Secondary Outcome: Mean Absolute Change From Baseline in Patient Oriented Eczema Measure (POEM)
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following POEM endpoints:
  • Mean absolute change from baseline in Patient Oriented Eczema Measure (POEM)
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

30. Secondary Outcome: Mean Percentage Change From Baseline in Patient Oriented Eczema Measure (POEM)
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following POEM endpoints:
  • Mean percentage change from baseline in Patient Oriented Eczema Measure (POEM)
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

31. Secondary Outcome: Percentage of Participants Achieving a Reduction of ≥4 in the POEM Score, of Those With a Score of ≥4 at Baseline
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following POEM endpoints:
  • Percentage of participants achieving a reduction of ≥4 in the POEM score, of those with a score of ≥4 at baseline
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

32. Secondary Outcome: Number of Courses Per Patient-year of Any Rescue Medication (Not Including Antibacterial Therapy)
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following Rescue therapy use endpoints:
  • Number of courses per patient-year of any rescue medication (not including antibacterial therapy)
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

33. Secondary Outcome: Number of Courses Per Patient-year of Topical Corticosteroids of Any Potency
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following Rescue therapy use endpoints:
  • Number of courses per patient-year of topical corticosteroids of any potency
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

34. Secondary Outcome: Number of Courses Per Patient-year of Topical Tacrolimus (0.1%), Topical Pimecrolimus (1%) or Grade VII Topical Corticosteroid
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following Rescue therapy use endpoints:
  • Number of courses per patient-year of topical tacrolimus (0.1%), topical pimecrolimus
  (1%) or grade VII topical corticosteroid
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

35. Secondary Outcome: Number of Courses Per Patient Year of Moderate Potency (Grade IV and V) Topical Steroids
Description: The efficacy of long-term treatment with EDP1815 in the treatment of Atopic Dermatitis will be measured using the following Rescue therapy use endpoints:
  • Number of courses per patient year of moderate potency (grade IV and V) topical steroids
Time Frame: 40 weeks
Population: as for outcome 1
Arm/Group | Group 1 | Group 2 | Group 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from informed consent, during the treatment period (110 days on average) and through an additional 28 days after taking their last dose of study drug.
Arm/Group | Group 1 | Group 2 | Group 3
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/102 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/104 | 1/102 | 1/79
Other Adverse Events (participants affected / at risk) | 26/104 | 20/102 | 5/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=104) | Group 2 (N=102) | Group 3 (N=79)
Hypertension Exacerbation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=104) | Group 2 (N=102) | Group 3 (N=79)
Nasopharyngitis (Infections and infestations) | 9 (12) | 6 (8) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 7 (10) | 3 (3)
COVID-19 (Infections and infestations) | 8 (8) | 3 (3) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 (12) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the study, the data may be considered for reporting at a scientific meeting or for publication in a scientific journal. The sponsor has final approved authority over publication of the study data.

DOCUMENTS (2):
  • Study Protocol (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/41/NCT05439941/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/41/NCT05439941/SAP_001.pdf